CLINICAL TRIAL: NCT04999761
Title: Platform Study of AB122 Based Treatments in Patients with Advanced Solid Tumors
Brief Title: AB122 Platform Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10071010
Record Dates: First submitted 2021-07-27; First posted 2021-08-11 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Advanced or Metastatic Solid Tumor; Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; Non-small Cell Lung Cancer; Gastric Cancer; Alveolar Soft Part Sarcoma; Esophageal Cancer; Head and Neck Cancer; Biliary Tract Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Sarcoma, Alveolar Soft Part; Esophageal Neoplasms; Head and Neck Neoplasms; Biliary Tract Neoplasms | interventions — TAS-116; futibatinib; 4-(2-fluoro-4-((((2-phenylacetyl)amino)thioxomethyl)amino)phenoxy)-7-methoxy-N-methyl-6-quinolinecarboxamide; trifluridine tipiracil drug combination; Ramucirumab; Bevacizumab; Fluorouracil; Cisplatin; Carboplatin; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (17):
- Cohort A-1 (Experimental): AB122 will be given in participants with advanced or metastatic solid tumor.
  Interventions: Drug: AB122
- Cohort A-2 (Experimental): AB122 will be given in participants with advanced or metastatic solid tumor.
  Interventions: Drug: AB122
- Cohort B-1 (Experimental): AB122 will be given in combination with TAS-116 in participants with pancreatic ductal adenocarcinoma.
  Interventions: Drug: AB122; Drug: TAS-116
- Cohort B-2 (Experimental): AB122 will be given in combination with TAS-116 in participants with unresectable metastatic MSS/pMMR CRC without liver metastases.
  Interventions: Drug: AB122; Drug: TAS-116
- Cohort B-3 (Experimental): AB122 will be given in combination with TAS-116 in participants with unresectable metastatic non-squamous NSCLC without actionable gene alterations.
  Interventions: Drug: AB122; Drug: TAS-116
- Cohort D-1 (Experimental): AB122 will be given in combination with TAS-120 in participants with unresectable metastatic NSCLC with PD-L1 high expression and without actionable gene alterations.
  Interventions: Drug: AB122; Drug: TAS-120
- Cohort E-1 (Experimental): AB122 will be given in combination with TAS-115 in participants with unresectable metastatic NSCLC without actionable gene alterations.
  Interventions: Drug: AB122; Drug: TAS-115
- Cohort E-2 (Experimental): AB122 will be given in combination with TAS-115 in participants with unresectable metastatic ASPS, in those who received or no prior regimen for advanced disease.
  Interventions: Drug: AB122; Drug: TAS-115
- Cohort C-1 (Experimental): AB122 will be given in combination with TAS-102 and Ramucirumab in participants with unresectable or recurrent gastric cancer or gastroesophageal junction cancer.
  Interventions: Drug: AB122; Drug: TAS-102; Drug: Ramucirumab
- Cohort C-2 (Experimental): AB122 will be given in combination with TAS-102 and Bevacizumab in participants with unresectable metastatic CRC.
  Interventions: Drug: AB122; Drug: TAS-102; Drug: Bevacizumab
- Cohort D-2 (Experimental): AB122 will be given in combination with TAS-120, Fluorouracil and Cisplatin in participants with histologically diagnosed advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus with no prior treatment for advanced cancer.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: Fluorouracil; Drug: Cisplatin
- Cohort D-3 (Experimental): AB122 will be given in combination with TAS-120 and AB154 in participants with histologically diagnosed advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus with no prior treatment for advanced cancer or who have been previously treated with one line of chemotherapy.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: AB154
- Cohort D-4 (Experimental): AB122 will be given in combination with TAS-120, Fluorouracil and Cisplatin/Carboplatin in participants with histologically diagnosed advanced or metastatic squamous cell carcinoma of the head and neck (middle pharynx, oral cavity, hypopharynx, larynx) with no prior treatment for advanced cancer.
  ・The validity of enrollment in the cohort must be confirmed, taking into account the patient background including CPS and the guidelines for head and neck cancer treatment.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: Fluorouracil; Drug: Carboplatin; Drug: Cisplatin
- Cohort D-5 (Experimental): AB122 will be given in combination with TAS-120 and AB154 in participants with histologically diagnosed advanced or metastatic squamous cell carcinoma of the head and neck (middle pharynx, oral cavity, hypopharynx, larynx) with no prior treatment for advanced cancer.
  ・The validity of enrollment in the cohort must be confirmed, taking into account the patient background including CPS and the guidelines for head and neck cancer treatment.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: AB154
- Cohort D-6 (Experimental): AB122 will be given in combination with TAS-120, Carboplatin and nab-Paclitaxel in participants with unresectable metastatic squamous NSCLC patients with no prior treatment for advanced cancer.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: Carboplatin; Drug: nab-Paclitaxel
- Cohort D-7 (Experimental): AB122 will be given in combination with TAS-120, Cisplatin and Gemcitabine in participants with unresectable metastatic adenocarcinoma or adenosquamous biliary tract cancer patients with no prior treatment for advanced cancer.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: Cisplatin; Drug: Gemcitabine
- Cohort D-8 (Experimental): AB122 will be given in combination with TAS-120, nab-Paclitaxel and Gemcitabine in participants with unresectable metastatic Pancreatic ductal adenocarcinoma patients with no prior treatment for advanced cancer.
  Interventions: Drug: AB122; Drug: TAS-120; Drug: nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes Q3W.
  Arms: Cohort A-2
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes Q2W.
  Arms: Cohort B-1
Drug: TAS-116 — TAS-116 will be administered orally in 5-day on and 2-day off schedule on an empty stomach at least 1 hour before or 2 hour after eating.
  Arms: Cohort B-1
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes Q2W.
  Arms: Cohort B-2
Drug: TAS-116 — TAS-116 will be administered orally in 5-day on and 2-day off schedule on an empty stomach at least 1 hour before or 2 hour after eating.
  Arms: Cohort B-2
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes Q2W.
  Arms: Cohort B-3
Drug: TAS-116 — TAS-116 will be administered orally in 5-day on and 2-day off schedule on an empty stomach at least 1 hour before or 2 hour after eating.
  Arms: Cohort B-3
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-1
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-1
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort E-1
Drug: TAS-115 — TAS-115 will be administered orally in 5-day on and 2-day off schedule on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort E-1
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort E-2
Drug: TAS-115 — TAS-115 will be administered orally in 5-day on and 2-day off schedule on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort E-2
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes every 2 weeks.
  Arms: Cohort C-1
Drug: TAS-102 — TAS-102 will be administered orally twice daily at a dose calculated based on body surface area (BSA) within 1 hour after morning and evening meals for 5 days, a week with 2 days rest for 2 weeks, followed by a 14-day rest, repeated every 4 weeks.
  Arms: Cohort C-1
Drug: Ramucirumab — Ramucirumab will be administered by infusion at a dose calculated using the body weight over approximately 60 minutes every 2 weeks.
  Arms: Cohort C-1
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes every 2 weeks.
  Arms: Cohort C-2
Drug: TAS-102 — TAS-102 will be administered orally twice daily at a dose calculated based on BSA within 1 hour after morning and evening meals for 5 days, a week with 2 days rest for 2 weeks, followed by a 14-day rest, repeated every 4 weeks.
  Arms: Cohort C-2
Drug: Bevacizumab — Bevacizumab will be administered by infusion at a dose calculated using the body weight over approximately 90 minutes every 2 weeks.
  Arms: Cohort C-2
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes Q2W.
  Arms: Cohort A-1
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-2
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-2
Drug: Fluorouracil — Fluorouracil will be administered with 800 mg/m2/day given by continuous intravenous infusion from Day 1 to Day 5.
  Arms: Cohort D-2
Drug: Cisplatin — Cisplatin will be administered with 80 mg/m2 given by infusion every 3 weeks.
  Arms: Cohort D-2
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-3
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-3
Drug: AB154 — AB154 will be administered with 1200 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-3
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-4
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-4
Drug: Fluorouracil — Fluorouracil will be administered with 1000 mg/m2/day given by continuous intravenous infusion from Day 1 to Day 4.
  Arms: Cohort D-4
Drug: Carboplatin — Carboplatin will be administered with AUC 5 given by infusion every 3 weeks.
  Arms: Cohort D-4
Drug: Cisplatin — Cisplatin will be administered with 100 mg/m2 given by infusion every 3 weeks.
  Arms: Cohort D-4
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-5
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-5
Drug: AB154 — AB154 will be administered with 1200 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-5
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-6
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-6
Drug: Carboplatin — Carboplatin will be administered with AUC 6 given by infusion every 3 weeks.
  Arms: Cohort D-6
Drug: nab-Paclitaxel — Nab-Paclitaxel will be administered with 100 mg/m2 given by infusion on Day 1, Day 8 and Day 15.
  Arms: Cohort D-6
Drug: AB122 — AB122 will be administered with 360 mg/body given by infusion over 60 minutes every 3 weeks.
  Arms: Cohort D-7
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-7
Drug: Cisplatin — Cisplatin will be administered with 25 mg/m2 given by infusion on Day 1 and Day 8.
  Arms: Cohort D-7
Drug: Gemcitabine — Gemcitabine will be administered with 1000 mg/m2 given by infusion on Day 1 and Day 8.
  Arms: Cohort D-7
Drug: AB122 — AB122 will be administered with 240 mg/body given by infusion over 60 minutes every 2 weeks.
  Arms: Cohort D-8
Drug: TAS-120 — TAS-120 will be administered orally once daily (QD) on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Cohort D-8
Drug: nab-Paclitaxel — Nab-Paclitaxel will be administered with 125 mg/m2 given by infusion on Day 1, Day 8 and Day 15.
  Arms: Cohort D-8
Drug: Gemcitabine — Gemcitabine will be administered with 1000 mg/m2 given by infusion on Day 1, Day 8 and Day 15.
  Arms: Cohort D-8

SUMMARY:
This is a phase 1, non-randomized open-label, multicenter platform study designed to evaluate the tolerability and safety of AB122 in patients with malignancies specified in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female aged ≥ 18 years at the time of informed consent; Willing and able to comply with scheduled visits and study procedures (except for Cohort E-2);
* Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 before administration of study treatment;
* Has adequate organ function as defined by the following criteria:

  * AST and ALT ≤ 3 × ULN; or if a patient with documented liver metastases, AST and ALT ≤ 5 × ULN
  * T-Bil of ≤ 1.5 × ULN
  * ANC ≥ 1500 /mm3 (ie, ≥ 1.5 × 109 /L by International System of Units [SI]) (excluding measurements obtained within 7 days after administration of granulocyte colony-stimulating factor [G-CSF])
  * Platelet count ≥ 100000 /mm3 (SI: ≥ 100 × 109 /L) (excluding measurements obtained within 7 days after a transfusion of platelets)
  * Hemoglobin value of ≥ 9.0 g/dL excluding measurements within 4 weeks after a transfusion of packed red blood cells (RBCs) or whole blood
* Has a life expectancy of at least 90 days;

Cohort A-1 and A-2

* Japanese male and female;
* Has a histologically or cytologically confirmed diagnosis of solid tumor;
* Has disease progression after standard treatment for advanced or metastatic disease, are intolerant to the standard treatment;

Cohort B-1

* Has a histologically or cytologically confirmed diagnosis of PDAC;
* Has disease progression after or intolerant to one prior systemic chemotherapy for advanced or metastatic disease

Cohort B-2

* Has a histologically or cytologically confirmed diagnosis of CRC.
* Has been received one regimen of standard chemotherapy for advanced or metastatic disease, and was refractory or intolerant to the chemotherapy

Cohort B-3 - Has a histologically or cytologically confirmed non-squamous NSCLC;

* Has been received one or two regimen of standard chemotherapy for advanced or metastatic disease, and was refractory or intolerant to the standard treatment
* Has been most recently received regimen including an ICI (anti PD-1 antibodies, anti PD-L1 antibodies or anti CTLA-4 antibodies) and platinum-based chemotherapy in combination or in sequence (i.e., platinum-based chemotherapy followed by checkpoint inhibitor therapy), and all of the following criteria must be met:

  * Received at least 2 doses at the most recent ICI therapy
  * Radiographic complete response or partial response based on investigator assessment with ICI therapy
  * Documented radiographic disease progression with above most recently received regimen

Cohort C-1

* Has unresectable advanced or recurrent gastric cancer or gastroesophageal junction cancer as pathologically confirmed adenocarcinoma
* Gastroesophageal junction cancer is defined as a tumor with an epicenter that is located within 2 cm proximal to and distal from the esophagogastric junction (the boundary of esophageal and gastric muscularis).
* Has received 2-4 standard regimens listed below and has demonstrated disease progression according to imaging test during the most recent treatment or within 12 weeks after the final dose (The patient is eligible if the treatment is discontinued owing to SAEs, allergic reactions, or neurotoxicities.):

  * fluoropyrimidines and platinum
  * taxane or irinotecan
  * ramucirumab

Cohort C-2

* Has histologically confirmed unresectable adenocarcinoma of the colon or rectum (all other histological types are excluded)
* RAS status must have been previously determined (mutant or wild-type) based on local assessment of tumor biopsy; Wild type is defined as v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) (exon 2, 3 and 4) and neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS) (exon 2, 3 and 4) wild type. [Mutant is defined as at least KRAS or NRAS mutant (any exon, any mutation)].
* Has received at least 2 prior chemotherapy regimens for the treatment of advanced CRC and had demonstrated disease progression according to imaging test during the most recent treatment or within 12 weeks after the final dose , or intolerance to their last regimen, and all of the following criteria must be met:

  * Prior treatment regimens must have included a fluoropyrimidine, irinotecan, oxaliplatin, an anti-VEGF monoclonal antibody
  * For RAS wild-type patients, an anti-EGFR monoclonal antibody must have included in addition to above

Cohort D-1

* Has histologically confirmed advanced or metastatic NSCLC regardless of histologic type.
* Has PD-L1 (≥ 50% tumor proportion score) in tumor tissue sample as determined at a local laboratory.

Cohort D-2

* Has histologically diagnosed advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus.
* No prior therapy for advanced or metastatic disease. • Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy.

Cohort D-3

* Has histologically diagnosed advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus.
* No prior therapy for advanced or metastatic disease, or refractory or intolerant to at least 1 cycle of standard first-line therapy.

  * Treatment discontinued due to intolerable toxicity or because the same drug cannot be re-treated before the disease progresses is considered as intolerable to the previous treatment.
  * Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy.

Cohort D-4

* Has histologically or cytologically confirmed recurrent or advanced squamous head and neck cancer (oropharynx, oral mucosa, hypopharynx, larynx).

  * The confirmed status of the human papillomavirus (HPV) in cancers of the mid-pharynx.
  * Patient background such as combined positive score (CPS) and head and neck cancer treatment guidelines must be taken into account to confirm the validity of enrollment in this cohort.
* No prior therapy for advanced or metastatic disease. • Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy. • Treatment of locally advanced disease completed more than 6 months prior to the start of study drug administration is not considered prior therapy.

Cohort D-5

* Has histologically or cytologically confirmed recurrent or advanced squamous head and neck cancer (oropharynx, oral mucosa, hypopharynx, larynx).

  * The confirmed status of the HPV in cancers of the mid-pharynx.
  * Patient background such as CPS and head and neck cancer treatment guidelines must be taken into account to confirm the validity of enrollment in this cohort.
* No prior therapy for advanced or metastatic disease. • Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy. • Treatment of locally advanced disease completed more than 6 months prior to the start of study drug administration is not considered prior therapy.

Cohort D-6

* Has histologically or cytologically confirmed recurrent or advanced squamous NSCLC.
* No prior therapy for advanced or metastatic disease. • Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy.

Cohort D-7

* Has histologically confirmed unresectable or advanced biliary tract cancer (intrahepatic bile duct, extrahepatic bile duct, gallbladder, or duodenal papillary region) with a diagnosis of adenocarcinoma or adenosquamous carcinoma.
* No prior therapy for advanced or metastatic disease. • Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy.

Cohort D-8

* Has histologically confirmed unresectable or advanced pancreatic ductal adenocarcinoma (highly differentiated, moderately differentiated, or poorly differentiated).
* No prior therapy for advanced or metastatic disease. Adjuvant therapy or neo adjuvant therapy is not considered as prior therapy if there is no recurrence during or within 6 months after completion of the therapy.

Cohort E-1

* Has a histologically or cytologically confirmed advanced or metastatic NSCLC regardless of histologic type.
* Has PD-L1 (≥ 50% tumor proportion score) in tumor tissue sample as determined at a local laboratory (except for tolerability part).
* Has been received 1-4 regimen for advanced or metastatic disease
* Has been received one regimen of ICI monotherapy or combination therapy (anti PD-1 antibodies, anti PD-L1 antibodies or anti CTLA-4 antibodies), and all of the following criteria must be met:

  * Received at least 2 doses of the ICI therapy
  * Documented radiographic disease progression with or after ICI therapy

Cohort E-2

* Has a histologically or cytologically confirmed advanced or metastatic ASPS
* Is male or female aged ≥ 16 years at the time of informed consent; Willing and able to comply with scheduled visits and study procedure

Exclusion Criteria:

* History or current evidence of cardiac arrhythmia and/or conduction abnormality: Any factor that can increase the risk of corrected QT interval (QTc) prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, etc.;
* Treatment with any of the following within the specified time frame prior to the day on which study treatment is scheduled to be started:

  * Major surgery within 4 weeks (the surgical incision should be fully healed prior to the day on which study treatment is scheduled to be started);
  * Extended-field radiotherapy within 4 weeks or limited-field radiotherapy within 2 weeks;
  * Any anticancer therapy within 2 weeks;
  * Any investigational agent received within 5 half-lives of the drug or 4 weeks, whichever shorter;
* Unresolved toxicity of ≥ Grade 2 attributed to any prior therapies (excluding anemia, peripheral sensory neuropathy, alopecia and skin pigmentation);
* A serious illness or medical condition(s) including, but not limited to, the following specific medical conditions:

  * Known acute systemic infection;
  * Known medical history of interstitial lung disease/ drug-induced interstitial lung disease/ radiation pneumonitis which required steroid treatment/ any evidence of clinically active interstitial lung disease;
  * Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV, Appendix A) within the previous 6 months; if > 6 months, cardiac function must be within normal limits and the patient must be free of cardiac-related symptoms;
  * Known severe chronic kidney disease;
  * Known positivity of human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody in baseline virus test. In addition, the patient who is known negative in HCV ribonucleic acid (RNA) is eligible, even if positive for HCV antibody;
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment, or may interfere with the interpretation of study results, and in the judgment of the investigator or sub-investigator would make the patient inappropriate for entry into this study;
* Previous or concurrent cancer that is distinct in primary disease or histology from the cancer being evaluated in this study, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (stage Ta, Tis and T1), cancers corresponding to intraepithelial or intramucosal neoplasia, or any cancer curatively treated > 5 years prior to the day on which study treatment is scheduled to be started;
* WOCBP or male patients who do not agree to effective birth control during the following period

  1. WOCBP patients: during the clinical study and until 100 days after the last dose of AB122, 180 days after TAS-116, TAS-102, TAS-120 or TAS-115, whichever is later;
  2. Male patients with WOCBP partners: during the clinical study and until 100 days after the last dose of AB122, 180 days after TAS-116, TAS-102, TAS-120 or TAS-115, whichever is later;
* Prior treatment with an anti-PD-L1 anti-PD-1, anti-CTLA-4, or other ICI or agonist as monotherapy or in combination (except for cohort B-3, C-1, D-1 tolerability part and E-1).
* Has received a live vaccine within 30 days prior to study treatment including, but not limited to the following examples: measles, mumps, rubella, varicella-zoster, yellow fever, and BCG. The inoculation with inactivated vaccines for seasonal influenza is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, ie, without evidence of progression for at least 28 days by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to enrollment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator. (eg, paresis of intestine, intestinal obstruction, unable to receive 5% dextrose in water [DW] in patients with diabetes mellitus, respiratory failure, renal failure, hepatic failure, cerebrovascular disorder, gastrointestinal ulcers that require transfusion or are hemorrhagic, and wounds/bone fractures associated with neovascularization during the healing process, accumulation of pleural within 2 weeks prior to enrollment, ascitic, or pericardial fluid requiring drainage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1a (All cohorts except Cohort D-4 and D-5) : Percentage of participants who experience a Dose Limiting Toxicity (DLT) | From first study treatment administration through Day 21 (Q3W arm) or Day 28 (Q2W arm)
Phase 1a (Cohort D-4 and D-5) : Percentage of adverse events and treatment-related adverse events. | From first study treatment administration through Day 21 (Q3W arm) or Day 28 (Q2W arm)
Phase 1b (Cohort B-n, D-n and E-n) : Objective Response Rate (ORR) | Through completion of treatment (estimated up to be 11 months)
Phase 1b (Cohort C-n): The 6-month PFS proportion by RECIST v1.1 | Through completion of treatment (estimated up to be 11 months)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (9):
- Japan (9):
  - A site selected by Taiho Pharmaceutical Co., Ltd., Aichi
  - A site selected by Taiho Pharmaceutical Co., Ltd., Chiba
  - A site selected by Taiho Pharmaceutical Co., Ltd., Ehime
  - A site selected by Taiho Pharmaceutical Co., Ltd., Hokkaido
  - A site selected by Taiho Pharmaceutical Co., Ltd., Kanagawa
  - A site selected by Taiho Pharmaceutical Co., Ltd., Osaka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Shizuoka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo
  - A site selected by Taiho Pharmaceutical Co., Ltd., Wakayama

IPD SHARING:
Plan to Share IPD: No
Data will not be shared according to the Sponsor policy on data sharing. Taiho policy on data sharing may be found at https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html.